CLINICAL TRIAL: NCT03773952
Title: A Phase IIa (Proof of Concept), Randomized, Double Blind, Placebo Controlled, Multicenter Clinical Trial to Evaluate the Safety and Efficacy of Oral Treatment With PBF-677 in Patients With Mild to Moderate Ulcerative Colitis
Brief Title: Safety and Efficacy of PBF-677 in Ulcerative Colitis Patients
Acronym: ADENOIBD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palobiofarma SL (Industry)
Collaborators: Qualitecfarma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBF-677-3
Record Dates: First submitted 2018-11-30; First posted 2018-12-12 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: randomized, double blind, placebo controlled, multicenter clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral 5-ASA + PBF-677 200 mg (Experimental): Oral Mesalazine (5-ASA) (4g) + PBF-677 (200mg)
  Interventions: Drug: PBF-677
- Oral 5-ASA + Placebo oral Capsules (Placebo Comparator): Oral Mesalazine (5-ASA) (4g) + Placebo oral capsules
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: PBF-677 — oral small molecule, antagonist of Adenosine A3 receptor (AA3R)
  Arms: Oral 5-ASA + PBF-677 200 mg
Drug: Placebo oral capsule — Oral capsules
  Arms: Oral 5-ASA + Placebo oral Capsules

SUMMARY:
This is a Phase IIa (proof of concept), randomized, double blind, placebo-controlled, multicentre clinical trial to evaluate the safety and efficacy of daily PBF-677 oral treatment during 28 days in Ulcerative colitis (UC) patients who are not receiving immunosuppressants and present mild-to-moderate activity of the disease. Enrolled patients would receive standard high doses of 5-ASA (4g), according to current clinical guidelines, and are randomized to receive also PBF-677 or placebo.

DETAILED DESCRIPTION:
This Proof-of-concept clinical trial is carefully designed to establish the safety profile of PBF-677 over 28 days in mild to moderate ulcerative colitis population and explore the relationship between the 200 mg PBF-677 dose and induction of remission, according to clinical parameters (Partial Mayo Score) and a faecal surrogate biomarker of mucosal inflammation (Calprotectin). The trial also will explore the PBF-677 pharmacokinetics (PK) profile during 28 days of administration.

This small-scale study has been designed to detect a signal that PBF-677 is safe and active on decreasing levels of faecal calprotectin, as well as preliminary evidence of ameliorate the Partial Mayo Clinical Score in colitis patients who are in flare of the disease.

The Population Under Study will be: Around 30 subjects. Adults (18-75 years old) non-immunosuppressed patients with mild to moderate active ulcerative colitis disease.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent
* Male or Female, 18 to 75 years of age, inclusive
* Patient with previous diagnosis of ulcerative colitis: ulcerative proctitis, left-side ulcerative colitis or extensive/pancolitis (E1, E2 and E3 of Montreal Classification, respectively) established at least 3 months prior to screening and determined by ordinary clinical, endoscopic, and histological procedures.
* Patient who has stable oral 5-ASA dose < 4 gr/day treatment, within 1 month prior to screening.
* Mild-to-moderate activity of the disease determined clinically during the screening period by Partial Mayo Clinical Score of ≤ 6, with rectal bleeding score ≤ 2 and/or a bowel frequency score ≤ 2.
* Patient in flare of the disease.
* Patient with faecal calprotectin levels > 50 mg/Kg
* Availability for the entire study period, absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; willingness to adhere to the protocol requirements, ability to cooperate adequately, to understand and follow the instructions of the physician or designee.
* Women who are not postmenopausal (at least 12 months) or surgically sterile must have a negative pregnancy test at screening and at the end of study and either abstain from sexual intercourse or use a highly effective method of birth control for the duration of the study and after 12 weeks after the last dose of study drug.
* For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm for the duration of the study and after 12 weeks from the last dose of study drug.

Exclusion Criteria:

* Patient who has treatment, within 3 months prior to screening, with immunomodulators including corticosteroids, azathioprine, mercaptopurine, biologics, tacrolimus, cyclosporine, for disease control.
* Patient who has stable oral 5-ASA dose ≥ 4 gr/day treatment, within 1 month prior to screening.
* Patient with C-reactive Protein levels (CRP) ≥ 10 mg/L
* Patient who has anti-diarrheal treatment, within 3 months prior to screening.
* Use of prescription medications started or with a dose adjustment within 4 weeks prior to study enrolment, or OTC medications or supplements started or with a dose adjustment within 2 weeks prior study enrolment.
* Use of products, food supplements or medical devices, whose composition includes probiotics in the 3 months prior to the selection.
* Patient who has fulminant or severe colitis, toxic megacolon, primary sclerosing cholangitis, Crohn's disease, history of colitis associated colonic dysplasia or active peptic ulcer disease.
* Patient who has prior extensive colonic resection, subtotal or total colectomy or planned surgery for UC
* Patient who has past or present fistula or abdominal abscess
* Patient who has clinically significant diseases and/or infections captured in the medical history or evidence of clinically significant findings on physical examination and/or clinically significant ordinary laboratory evaluations (haematology, biochemistry, and urinalysis) or ECG.
* Patient who has evidence of significant liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
* Patient who is currently participating in another clinical trial of an investigational drug or medical device within 90 days prior to screening.
* Patient who is pregnant or lactating
* Inability to comply with study protocol, in opinion of the investigator
* History of alcohol, drug or chemical abuse within 6 months prior to screening
* History of cancer except local basal or squamous cell carcinoma of the skin that has been excised and is considered cured.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-related adverse events as assessed by CTCAE v4.03" | 28 Days
  Adverse events will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. If

SECONDARY OUTCOMES:
Effect of PBF-677 on Faecal calprotectin levels | 28 Days
  Calprotectin levels in stools is a validated biomarker of the severity of the disease. A decrease in the calprotectin levels under 50 mg/Kg is associated with the remission of the disease flare.
Effect of PBF-677 on Ulcerative Colitis activity | 28 Days
  The assessment Will be based on the Partial Mayo Scoring Index that sum and score the following ítems:
  1. Stool Frequency (based on the past 3 days)
  2. Rectal Bleeding (based on the past 3 days)
  3. Physician's Global Assessment
  The scoring range is as follow:
  Remission = 0-1 Mild Disease = 2-4 Moderate Disease = 5-6 Severe Disease =7-9
Pharmacokinetic PBF-677 peak concentration in plasma | Day 1 and Day 14
  The parameter will be calculated from plasma samples collected at days 1 and 14 after drug administration. It will consist in the maximum plasma concentration (ng/mL) of PBF-677 observed after administration
Pharmacokinetic Time to PBF-677 peak concentration in plasma "Tmax" | Day 1 and Day 14
  The parameter will be calculated from plasma samples collected at days 1 and 14 after drug administration.It will consist in the time (in minutes) to reach the maximum "PBF-677" concentration in plasma samples of patients after oral administration of PBF-677.
Pharmacokinetic Area under curve (AUC) of PBF-677 in plasma | Day 1 and Day 14
  The parameter will be calculated from plasma samples collected at days 1 and 14 after drug administration. It will consist in the area under the concentration-time curve from zero up to ∞ with extrapolation of the terminal phase. "AUC(0-inf)" will be given in Amount·time/ volume units
Pharmacokinetic Ctrough plasma concentration of PBF-677 | Day 1 and Day 14
  Trough plasma concentration (measured concentration at the end of a dosing interval at steady state [taken directly before next administration])

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Enfermedad Inflamatoria Intestinal / IBD Unit. Servicio de Gastroenterología y Hepatología / Gastroenterology and Hepatology Dpt. Study Medical Coordinator Hospital Universitario Puerta de Hierro, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No